CLINICAL TRIAL: NCT01624233
Title: A Multicenter, Open-Label, Long-Term Study to Evaluate the Efficacy and Safety of LY2439821 in Japanese Patients With Moderate-to-Severe Psoriasis
Brief Title: A Study in Japanese Participants With Moderate-to-Severe Psoriasis
Acronym: UNCOVER-J
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13976; I1F-JE-RHAT (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-06-18; First posted 2012-06-20 (Estimated); Results first posted 2016-09-30 (Estimated); Last update posted 2019-09-10 (Actual); Status verified 2019-08

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — ixekizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 80 mg ixekizumab (Experimental): Administered by two 80 milligram (mg) subcutaneous (SC) injections at Week 0, followed by one 80 mg SC injection per Dosing Regimen 1 up to Week 12. Then administered by one 80 mg SC injection per Dosing Regimen 2 from Week 12 up to Week 52, and for up to 192 weeks following disease relapse occurring during a drug-free period beyond 52 weeks.
  Interventions: Drug: 80 mg ixekizumab

INTERVENTIONS:
Drug: 80 mg ixekizumab — Administered SC
  Other Names: LY2439821

SUMMARY:
This study will assess the safety and efficacy of ixekizumab in participants with moderate to severe psoriasis in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Men must agree to use a reliable method of birth control during the study
* Women must agree to use birth control or remain abstinent during the study and for at least 12 weeks after stopping treatment
* Candidates for phototherapy and/or systemic therapy
* Present with chronic psoriasis based on a confirmed psoriasis diagnosis for at least 6 months prior to enrollment
* At least 10% Body Surface Area (BSA) of Psoriasis at screening and at enrollment for participants with plaque psoriasis
* Static Physician Global Assessment (sPGA) score of at least 3 and Psoriasis Area and Severity Index (PASI) score of at least 12 at screening and at enrollment for participants with plaque psoriasis

Exclusion Criteria:

* History of drug-induced psoriasis
* Concurrent or recent use of any biologic agent
* Received systemic psoriasis therapy [such as psoralen and ultraviolet A (PUVA) light therapy] or phototherapy within the previous 4 weeks; or had topical psoriasis treatment within the previous 2 weeks prior to enrollment for participants with plaque psoriasis
* Cannot avoid excessive sun exposure or use of tanning booths for at least 4 weeks prior to enrollment and during the study
* Have participated in any study with interleukin-17(IL-17) antagonists, including ixekizumab
* Serious disorder or illness other than psoriasis
* Serious infection within the last 3 months
* Breastfeeding or nursing (lactating) women
* Clinically significant flare of psoriasis during the 12 weeks prior to enrollment for participants with plaque psoriasis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2012-06; Primary Completion 2013-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (17):
- Japan (17):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ehime
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gifu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ishikawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kumamoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miyazaki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Numakunai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Okayama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka-Pref
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saitama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Honma M, Cai Z, Burge R, Zhu B, Yotsukura S, Torisu-Itakura H. Relationship Between Rapid Skin Clearance and Quality of Life Benefit: Post Hoc Analysis of Japanese Patients with Moderate-to-Severe Psoriasis Treated with Ixekizumab (UNCOVER-J). Dermatol Ther (Heidelb). 2020 Dec;10(6):1397-1404. doi: 10.1007/s13555-020-00441-4. Epub 2020 Sep 10. PMID 32910360
- [Derived] Saeki H, Nakagawa H, Ishii T, Morisaki Y, Aoki T, Berclaz PY, Heffernan M. Efficacy and safety of open-label ixekizumab treatment in Japanese patients with moderate-to-severe plaque psoriasis, erythrodermic psoriasis and generalized pustular psoriasis. J Eur Acad Dermatol Venereol. 2015 Jun;29(6):1148-55. doi: 10.1111/jdv.12773. Epub 2014 Oct 30. PMID 25355284

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Period 2-Induction Dosing Period (Weeks 0 up to 12), Period 3-Maintenance Dosing Period (Weeks 12 up to 52), Period 4-Drug Free Period (Weeks 52 up to 100), Period 5-Retreatment Period (up to 192 additional weeks) and Period 6-Post-Treatment Follow-Up Period up to 12 weeks after the last visit.
Groups:
- 80 mg Ixekizumab (LY2439821): Ixekizumab:
  Period 2 - Participants were administered two 80-milligram (mg) subcutaneous (SC) injections at Week 0, followed by 80 mg given as 1 SC injection every 2 weeks (Q2W) (Weeks 2, 4, 6, 8, and 10).
  Period 3 - Participants were administered 80-mg as 1 SC injection every 4 weeks (Q4W) (Week 12 up to Week 52).
  Period 4 - No ixekizumab administered (drug-free). Period 5 - Participants who had a Ps relapse during the drug-free period (Period 4) or who completed Period 4 were administered 80-mg as 1 SC injection Q4W for up to 192 weeks.
Period: Period 2 - Induction
Arm/Group | 80 mg Ixekizumab (LY2439821)
Started | 91
Received at Least 1 Dose of Study Drug | 91
Erythrodermic Psoriasis (Ps) | 8
Pustular Ps | 5
Plaque Ps | 78
Completed | 90
Not Completed | 1
Not completed — Adverse Event | 1
Period: Period 3 - Maintenance
Arm/Group | 80 mg Ixekizumab (LY2439821)
Started | 90
Received at Least 1 Dose of Study Drug | 90
Completed | 83
Not Completed | 7
Not completed — Adverse Event | 2
Not completed — Lack of Efficacy | 1
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 2
Period: Period 4 - Drug Free Period
Arm/Group | 80 mg Ixekizumab (LY2439821)
Started | 70 (Only responders in participants with plaque Ps moved to the Drug Free Period 4.)
Adverse Event | 1 (1 participant who discontinued due to adverse event is included in the participants who relapsed.)
Physician Decision | 1 (1 participant who discontinued due to physician decision is included in the participants relapsed.)
Completed | 9
Not Completed | 61
Not completed — Relapsed | 61
Period: Period 5 - Retreatment Period
Arm/Group | 80 mg Ixekizumab (LY2439821)
Started | 80 (Period 5 included (participants with erythrodermic Ps or pustular Ps) or Period 4 completers.)
Completed | 70
Not Completed | 10
Not completed — Adverse Event | 5
Not completed — Lack of Efficacy | 1
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 3
Period: Period 6: Follow-up
Arm/Group | 80 mg Ixekizumab (LY2439821)
Started | 88 (Period 6 included participants received a dose of drug and exhibited the required neutrophil count.)
Completed | 79
Not Completed | 9
Not completed — Adverse Event | 3
Not completed — Lack of Efficacy | 2
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- 80 mg Ixekizumab (LY2439821): Ixekizumab:
  Period 2 - Participants were administered two 80-mg SC injections at Week 0, followed by 80-mg given as 1 SC injection Q2W (Weeks 2, 4, 6, 8, and 10).
  Period 3 - Participants were administered 80-mg as 1 SC injection Q4W (Week 12 up to Week 52) Period 4 - No ixekizumab administered (drug-free), (Week 52 up to Week 100) Period 5 - Participants who had a Ps relapse during the drug-free period (Period 4) or who completed Period 4 were administered 80 mg as 1 SC injection Q4W for up to 192 weeks.
Arm/Group | 80 mg Ixekizumab (LY2439821)
Number analyzed (Participants) | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (11.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 91
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 91
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Japan | 91
Psoriasis Area and Severity Index (PASI) Total Score [Mean (Standard Deviation); unit: units on a scale] — The PASI combines the extent of body surface involvement in 4 anatomical regions (head, trunk, arms, and legs). For each region the percent area of skin involved was estimated from 0 (0%) to 6 (90%-100%) and severity was estimated by clinical signs of erythema, induration and scaling with a scores range from 0(no involvement) to 4 (severe involvement). Each area is scored by itself and the scores were then combined for the final PASI. Overall scores range from 0 (no Ps) to 72 (the most severe disease).
  units on a scale | 27.24 (10.545)
Static Physician Global Assessment (sPGA) Score [Number; unit: participants] — The sPGA is the physician's determination of the participant's Ps lesions overall at a given time point. Lesions were categorized by descriptions for induration, erythema, and scaling. Participants Ps were assessed as clear (0), minimal (1), mild (2), moderate (3), severe (4), or very severe (5).
  participants
    0: Clear | 0
    1: Minimal | 0
    2: Mild | 1
    3: Moderate | 26
    4: Severe | 53
    5: Very Severe | 11
Percentage (%) of Body Surface Area (BSA) [Mean (Standard Deviation); unit: units on a scale] — BSA is a physician rating of the percentage of involvement of Ps for each participant. BSA is assessed on a continuous scale from 0% (no involvement) to 100% (full involvement), where 1% corresponds to the size of the participant's hand (includes the palm, fingers and thumb). Total BSA is the sum of handprints from the affected areas.
  units on a scale | 45.5 (23.22)
Nail Psoriasis Severity Index (NAPSI) Total Score [Mean (Standard Deviation); unit: units on a scale] — The NAPSI scale evaluates Ps severity in the fingernail bed and fingernail matrix with each divided into quadrants. Scores range from 0 (none) to 4 (Ps in all 4 quadrants), depending on the presence (score of 1) or absence (score of 0) of Ps in each quadrant of the fingernail bed or matrix. NAPSI score of a fingernail is the sum of scores from each quadrant of the fingernail bed and fingernail matrix (maximum of 8). The total NAPSI score equals the sum of all fingernails and ranges from 0 to 80. Higher scores indicate more severe Ps. Population: Only participants with non-missing data were included.
  units on a scale
    number analyzed (Participants) | 56
    (all) | 31.1 (22.16)
Psoriasis Scalp Severity Index (PSSI) Total Score [Mean (Standard Deviation); unit: units on a scale] — The PSSI is a physician assessment of erythema, induration and desquamation and percent of scalp that is covered with a scores range from 0 (none) to 4 (very severe). The composite score is derived from the sum of scores for erythema, induration, and desquamation multiplied by the score recorded for the extent of the scalp area involved, 1 (<10%) to 6 (90%-100%) with a total score ranging from 0 (less severity) to 72 (more severity). Population: Only participants with non-missing data were included.
  units on a scale
    number analyzed (Participants) | 87
    (all) | 27.0 (15.99)
Quick Inventory of Depressive Symptomatology-Self Reported 16 Items(QIDS-SR16) Total Score [Mean (Standard Deviation); unit: units on a scale] — QIDS-SR16 is a participant-administered, 16-item instrument assesses the existence and severity of symptoms of depression. A participant is asked a statement relating to the way they have felt for the past 7 days and rate on a 4-point scale: 0 (best) to 3 (worst). The sum of the domains [sad mood, concentration, self-criticism, suicidal ideation, interest, energy/fatigue, sleep disturbance, decrease/increase in appetite/weight, and psychomotor agitation/retardation] to give a single total scores range from 0 to 27, with higher scores indicating greater symptom severity.
  units on a scale | 4.6 (4.14)
Itch Numeric Rating Scale (NRS) Score [Mean (Standard Deviation); unit: units on a scale] — The Itch NRS is a participant-administered, 11-point horizontal scale anchored at 0 (no itch) and 10 (worst itch imaginable). Overall severity of a participant's itching from Ps is indicated by circling the number that best describes the worst level of itching in the past 24 hours.
  units on a scale | 6.1 (2.53)
Quick Inventory of Depressive Symptomatology-Self Reported (DLQI) Total Score [Mean (Standard Deviation); unit: units on a scale] — DLQI is a participant-administered, 10-question, validated, quality-of-life questionnaire that covers 6 domains, including symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. Response categories include 0 (not at all), 1 (a little), 2 (a lot), and 3 (very much) and unanswered ("not relevant") responses were scored as "0." Total scores range from 0 to 30, with higher score indicating greater quality of life impairment.
  units on a scale | 10.8 (6.50)
Joint Pain Visual Analog Scale (VAS) [Mean (Standard Deviation); unit: units on a scale] — The pain VAS is a participant-administered single-item scale designed to measure current joint pain from PsA using a 100-mm horizontal VAS. Overall severity of participant's joint pain from PsA is indicated by placing a single mark on the horizontal 100-mm scale from 0 mm (no pain) to 100 mm (pain as severe as you can imagine). Population: Only participants with non-missing data were included.
  units on a scale
    number analyzed (Participants) | 11
    (all) | 62.4 (23.79)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving ≥75% Improvement in Psoriasis Area and Severity Index (PASI) (Efficacy of Ixekizumab in Participants With Moderate to Severe Plaque Psoriasis. Measure: PASI)
Description: The PASI combines the extent of body surface involvement in 4 anatomical regions (head, trunk, arms, and legs). For each region the percent area of skin involved was estimated from 0 (0%) to 6 (90%-100%) and severity was estimated by clinical signs of erythema, induration and scaling with a scores range from 0 (no involvement) to 4 (severe involvement). Each area is scored by itself and the scores were then combined for the final PASI. Final PASI=sum of severity parameters for each region * area score * weighing factor [head (0.1), upper limbs (0.2), trunk (0.3), lower limbs (0.4)]. Overall scores range from 0 (no Ps) to 72 (the most severe disease).
Time Frame: Week (Wk) 12
Population: All participants with Plaque Ps who received at least one dose of study drug and had at least 1 measurement of PASI after study treatment. Non-responders and participants who discontinued at any time prior to specified time points were defined as non-responders for Non-Responder Imputation (NRI) analysis.
Measure: Number; unit: percentage of participants
Arm/Group | 80 mg Ixekizumab (LY2439821)
Number analyzed (Participants) | 78
percentage of participants | 98.7

2. Secondary Outcome: Percentage of Participants Achieving ≥75% Improvement in PASI
Description: The PASI combines the extent of body surface involvement in 4 anatomical regions (head, trunk, arms, and legs). For each region, the percent area of skin involved was estimated from 0 (0%) to 6 (90%-100%) and severity was estimated by clinical signs of erythema, induration and scaling with a scores range from 0 (no involvement) to 4 (severe involvement). Each area is scored by itself and the scores were then combined for the final PASI. Final PASI=sum of severity parameters for each region * area score * weighing factor [head (0.1), upper limbs (0.2), trunk (0.3), lower limbs (0.4)]. Overall scores range from 0 (no Ps) to 72 (the most severe disease).
Time Frame: Wks 24 and 52
Population: All participants with Plaque Ps who received at least 1 dose of study drug and had at least 1 measurement of PASI after study treatment. Non-responders and participants who discontinued at any time prior to Wk 52 were defined as non-responders for NRI analysis.
Measure: Number; unit: percentage of participants
Arm/Group | 80 mg Ixekizumab (LY2439821)
Number analyzed (Participants) | 78
percentage of participants
  Wk 24 | 95.9
  Wk 52 | 92.3

3. Secondary Outcome: Pharmacokinetics (PK): Ctrough at Steady State (Ctrough ss) of Ixekizumab
Description: PK samples were from 1 or 2 sampling cohorts. Ctrough is the minimum observed concentration of ixekizumab at steady state. Steady-state ixekizumab trough concentrations were summarized for the induction dosing period at week 12, the time of the primary efficacy assessment. Steady-state ixekizumab trough concentrations were summarized for the maintenance dosing period at week 24.
Time Frame: Pre-dose at Wks 12 (Day 84) and Wks24 (Day 168)
Population: All participants with Plaque Ps, Pustular Ps or Erythrodermic Ps who had at least 1 dose of study drug and evaluable Ctrough data at the specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/milliliter (µg/mL)
Arm/Group | 80 mg Ixekizumab (LY2439821)
Number analyzed (Participants) | 43
micrograms/milliliter (µg/mL)
  Wk 12 (80 mg Q2W) Cohort 2: number analyzed (Participants) | 22
  Wk 12 (80 mg Q2W) Cohort 2 | 9.63 (43.6)
  Wk 24 (80 mg Q4W) Cohort 1: number analyzed (Participants) | 21
  Wk 24 (80 mg Q4W) Cohort 1 | 3.48 (65.4)

4. Secondary Outcome: Number of Participants With Anti-Ixekizumab Antibodies
Description: Treatment-emergent immunogenicity is defined as any occurrence of a 4-fold or 2-dilution increase in titer over the pretreatment baseline titer. In the case of a negative result at baseline, treatment-emergent immunogenicity is defined as an increase in titer to ≥1:10.
Time Frame: Baseline through Wk 52
Population: All participants with Plaque Ps, Pustular Ps or Erythrodermic Ps who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | 80 mg Ixekizumab (LY2439821)
Number analyzed (Participants) | 91
participants
  Plaque Ps: number analyzed (Participants) | 78
  Plaque Ps | 10
  Erythrodermic Ps: number analyzed (Participants) | 8
  Erythrodermic Ps | 0
  Pustular Ps: number analyzed (Participants) | 5
  Pustular Ps | 0

5. Secondary Outcome: Percent of Participants Achieving PASI 90% and 100% Improvement
Description: as for outcome 1
Time Frame: Wks 12, 24 and 52
Population: All participants with Plaque Ps who received at least 1 dose of study drug and had at least 1 post-dose measurement of PASI after study treatment. Participants who discontinued treatment at any time prior to the specified time points were defined as non-responders for NRI at Wks 12 and 52.
Measure: Number; unit: percentage of participants
Arm/Group | 80 mg Ixekizumab (LY2439821)
Number analyzed (Participants) | 78
percentage of participants
  Wk 12 (80 mg Q2W) PASI 90% | 83.3
  Wk 12 (80 mg Q2W) PASI 100% | 32.1
  Wk 24 (80 mg Q4W) PASI 90% | 90.5
  Wk 24 (80 mg Q4W) PASI 100% | 48.6
  Wk 52 (80 mg Q4W) PASI 90% | 80.8
  Wk 52 (80 mg Q4W) PASI 100% | 48.7

6. Secondary Outcome: Percentage of Participants With Static Physician Global Assessment (sPGA) (0 or 1) or sPGA (0) (Efficacy of Ixekizumab in Participants With Moderate to Severe Plaque Psoriasis Measure: sPGA)
Description: The sPGA is the physician's determination of the participant's Ps lesions overall at a given time point. Lesions were categorized by descriptions for induration, erythema, and scaling. Participants Ps were assessed as 0 (clear) or 1 (minimal).
Time Frame: Wks 12, 24 and 52
Population: All participants with Plaque Ps who received at least 1 dose of study drug and had at least 1 post-dose measurement of sPGA after study treatment. Participants who discontinued treatment at any time prior to the specified time points were defined as non-responders for NRI analysis for Wks 12 and 52.
Measure: Number; unit: percentage of participants
Arm/Group | 80 mg Ixekizumab (LY2439821)
Number analyzed (Participants) | 78
percentage of participants
  Wk 12 (80 mg Q2W) sPGA (0 or 1) | 89.7
  Wk 24 (80 mg Q4W) sPGA (0 or 1) | 89.2
  Wk 52 (80 mg Q4W) sPGA (0 or 1) | 83.3
  Wk 12 (80 mg Q2W) sPGA (0) | 35.9
  Wk 24 (80 mg Q4W) sPGA (0) | 51.4
  Wk 52 (80 mg Q4W) sPGA (0) | 52.6

7. Secondary Outcome: Change From Baseline in Percent of Body Surface Area (BSA) Involvement
Description: BSA is a physician rating of the percentage of involvement of Ps for each participant. BSA is assessed on a continuous scale from 0% (no involvement) to 100% (full involvement), in which 1% corresponds to the size of the participants hand (includes the palm, fingers and thumb).
Time Frame: Baseline, Wk 12; Baseline, Wk 24; Baseline, Wk 52
Population: All participants with Plaque Ps with a baseline and at least 1 post-dose result. Participants with missing BSA at Wks 12 and 52 were imputed by last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: percentage of BSA
Arm/Group | 80 mg Ixekizumab (LY2439821)
Number analyzed (Participants) | 78
percentage of BSA
  Wk 12 (80 mg Q2W) | -38.3 (19.26)
  Wk 24 (80 mg Q4W) | -41.2 (20.23)
  Wk 52 (80 mg Q4W) | -40.8 (19.73)

8. Secondary Outcome: Change From Baseline in Nail Psoriasis Severity Index (NAPSI)
Description: The NAPSI is a numeric, reproducible, objective tool for evaluation of fingernail Ps. This scale is used to evaluate the severity of fingernail bed Ps and fingernail matrix Ps by area of involvement in the fingernail unit. The fingernail is divided with imaginary horizontal and longitudinal lines into quadrants. Each fingernail is given a score for fingernail bed Ps 0 (none) to 4 (Ps in 4 quadrants of the fingernail) and fingernail matrix Ps 0 (none) to 4 (Ps in 4 quadrants in matrix), depending on the presence (score of 1) or absence (score of 0) of any of the features of fingernail bed or matrix Ps in each quadrant. The NAPSI score of a fingernail is the sum of scores in fingernail bed and fingernail matrix from each quadrant (maximum of 8). Each fingernail is evaluated, then the sum of all fingernails equals the total NAPSI score with a range from range 0 to 80. Higher scores indicated more severe psoriasis.
Time Frame: Baseline, Wk 12; Baseline, Wk 24; Baseline, Wk 52
Population: All participants Plaque Ps with NAPSI at baseline and at least 1 post dose result. Participants with missing NAPSI at Wks 12 and 52 were imputed by LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 80 mg Ixekizumab (LY2439821)
Number analyzed (Participants) | 44
units on a scale
  Wk 12 (80 mg Q2W) | -7.7 (14.65)
  Wk 24 (80 mg Q4W) | -20.5 (19.42)
  Wk 52 (80 mg Q4W) | -23.4 (23.67)

9. Secondary Outcome: Change From Baseline in Psoriasis Scalp Severity Index (PSSI)
Description: The PSSI is a physician assessment of erythema, induration and desquamation and percent of scalp that is covered with a scores range from 0 (none) to 4 (very severe). The composite score is derived from the sum of scores for erythema, induration, and desquamation multiplied by the score recorded for the extent of the scalp area involved, 1 (<10%) to 6 (90%-100%) with a total scores range from 0 to 72, with lower scores indicating less severity.
Time Frame: Baseline, Wk 12; Baseline, Wk 24; Baseline, Wk 52
Population: All participants with Plaque Ps with a PSSI baseline and at least 1 post-dose result. Participants with missing PSSI at Wks 12 and 52 were imputed by LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 80 mg Ixekizumab (LY2439821)
Number analyzed (Participants) | 76
units on a scale
  Wk 12 (80 mg Q2W) | -24.8 (15.12)
  Wk 24 (80 mg Q4W) | -24.9 (15.11)
  Wk 52 (80 mg Q4W) | -23.3 (16.48)

10. Secondary Outcome: Change From Baseline in Quick Inventory of Depressive Symptomatology-Self Reported 16 Items (QIDS-SR16) Score [Quality of Life and Outcome Assessments. Measures: Patient Reported Outcomes (PRO)]
Description: QIDS-SR16 is a participant-administered, 16-item instrument intended to assess the existence and severity of symptoms of depression. A participant is asked to consider each statement as it relates to the way they have felt for the past 7 days and rate each on a 4-point scale: 0 (best) to 3 (worst). The sum of the 16 items corresponding to 9 depression domains [sad mood, concentration, self-criticism, suicidal ideation, interest, energy/fatigue, sleep disturbance (initial, middle and late insomnia or hypersomnia), decrease/increase in appetite/weight, and psychomotor agitation/retardation] to give a single total scores range from 0 to 27, with higher scores indicating greater symptom severity.
Time Frame: Baseline, Wk 12; Baseline, Wk 24; Baseline, Wk 52
Population: Participants with Plaque Ps who had QIDS-SR16 at baseline and at least 1 post-dose result. Participants with missing QIDS-SR16 at Wks 12 and 52 were imputed by LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 80 mg Ixekizumab (LY2439821)
Number analyzed (Participants) | 78
units on a scale
  Wk 12 (80 mg Q2W) | -1.1 (3.65)
  Wk 24 (80 mg Q4W) | -1.6 (3.80)
  Wk 52 (80 mg Q4W) | -1.4 (3.57)

11. Secondary Outcome: Change From Baseline in Itch Numeric Rating Scale (NRS) Score
Description: The Itch NRS is a participant-administered, 11-point horizontal scale anchored at 0 (no itch) and 10 (worst itch imaginable). Overall severity of a participant's itching from Ps is indicated by circling the number that best describes the worst level of itching in the past 24 hours.
Time Frame: Baseline, Wk 12; Baseline, Wk 24; Baseline, Wk 52
Population: Participants with Plaque Ps who had Itch NRS at baseline and at least 1 post-dose result. Participants with missing Itch NRS at Wks 12 and 52 were imputed by LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 80 mg Ixekizumab (LY2439821)
Number analyzed (Participants) | 78
units on a scale
  Wk 12 (80 mg Q2W) | -4.7 (2.68)
  Wk 24 (80 mg Q4W) | -4.8 (2.90)
  Wk 52 (80 mg Q4W) | -4.8 (2.83)

12. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Score
Description: DLQI is a participant-administered, 10-question, validated, quality-of-life questionnaire that covers 6 domains, including symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. Response categories include 0 (not at all), 1 (a little), 2 (a lot), and 3 (very much) and unanswered ("not relevant") responses were scored as "0." Total scores range from 0 to 30, with higher score indicating greater quality of life is impairment. A 5-point increase in total score from baseline is considered clinically relevant.
Time Frame: Baseline, Wk 12; Baseline, Wk 24; Baseline, Wk 52
Population: Participants with Plaques Ps who had DLQI at baseline and at least 1 post-dose result. Participants with missing DLQI at Wks 12 and 52 were imputed by LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 80 mg Ixekizumab (LY2439821)
Number analyzed (Participants) | 78
units on a scale
  Wk 12 (80 mg Q2W) | -9.2 (5.75)
  Wk 24 (80 mg Q4W) | -9.2 (6.57)
  Wk 52 (80 mg Q4W) | -9.6 (6.24)

13. Secondary Outcome: Number of Participants Achieving American College of Rheumatology 20% (ACR20) Improvement [Efficacy of Ixekizumab in Participants With Psoriatic Arthritis (PsA) as Measured by ACR20]
Description: ACR20 response is defined as a ≥20% improvement from baseline for tender joint count (TJC) and swollen joint count (SJC) and in at least 3 of the following 5 criteria: participant's assessment of Joint Pain visual analog scale (VAS), Patient's Global Assessment of Disease Activity VAS, Physician's Global Assessment of the Disease Activity VAS, participant's assessment of physical function using the Health Assessment Questionnaire Disability Index (HAQ-DI), or C-reactive protein (CRP) or the erythrocyte sedimentation rate (ESR).
Time Frame: Wks 12, 24 and 52
Population: Participants with PsA who had 3 or more tender joints and 3 or more swollen joints at screening and baseline.
Measure: Number; unit: participants
Arm/Group | 80 mg Ixekizumab (LY2439821)
Number analyzed (Participants) | 5
participants
  Wk 12 (80 mg Q2W) | 4
  Wk 24 (80 mg Q4W) | 4
  Wk 52 (80 mg Q4W) | 5

14. Secondary Outcome: Change From Baseline in Participants Assessment of Joint Pain Visual Analog Scale (VAS) (Efficacy of Ixekizumab in Participants With PsA Pain VAS)
Description: The pain VAS is a participant-administered single-item scale designed to measure current joint pain from PsA using a 100-mm horizontal VAS. Overall severity of participant's joint pain from PsA is indicated by placing a single mark on the horizontal 100-mm scale from 0 mm (no pain) to 100 mm (pain as severe as you can imagine).
Time Frame: Baseline, Wk 12; Baseline, Wk 52
Population: Participants with PsA who had 3 or more tender joints and 3 or more swollen joints at screening and baseline.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 80 mg Ixekizumab (LY2439821)
Number analyzed (Participants) | 5
mm
  Wk 12 (80 mg Q2W) | -47.3 (22.05)
  Wk 52 (80 mg Q4W) | -51.0 (19.05)

15. Secondary Outcome: Percent of Participants Achieving PASI 75%, 90% and/or 100% Improvement
Description: The PASI combines the extent of body surface involvement in 4 anatomical regions (head, trunk, arms, and legs). For each region the percent area of skin involved was estimated: 0 (0%) to 6 (90%-100%) and severity was estimated by clinical signs of erythema, induration and scaling, with a scores range from 0 (no involvement) to 4 (severe involvement). Each area is scored by itself and the scores were then combined for the final PASI. Final PASI=sum of severity parameters for each region * area score * weighing factor [head (0.1), upper limbs (0.2), trunk (0.3), lower limbs (0.4)]. Overall scores range from 0 (no Ps) to 72 (the most severe disease).
Time Frame: Wk 100 and Retreatment Wk 192
Population: All participants with Plaque Ps who received at least 1 dose of study drug and had at least 1 post-dose measurement of PASI after study treatment and entered Period 5. Participants who discontinued treatment at any time prior to the specified time points were defined as non-responders for NRI at Wks 100 and 192.
Measure: Number; unit: percentage of participants
Arm/Group | 80 mg Ixekizumab (LY2439821)
Number analyzed (Participants) | 67
percentage of participants
  Wk 100, PASI 75 | 7.5
  Wk 100, PASI 90 | 3.0
  Wk 100, PASI 100 | 0
  Wk 192, PASI 75 | 0
  Wk 192, PASI 90 | 0
  Wk 192, PASI 100 | 0

16. Secondary Outcome: Percentage of Participants With sPGA (0 or 1) and sPGA (0)
Description: as for outcome 6
Time Frame: Wk 100 and Retreatment Wk 192
Population: as for outcome 15
Measure: Number; unit: percentage of participants
Arm/Group | 80 mg Ixekizumab (LY2439821)
Number analyzed (Participants) | 67
percentage of participants
  Wk 100, sPGA(0, 1) | 4.5
  Wk 100, sPGA(0) | 0
  Wk 192, sPGA(0, 1) | 0
  Wk 192, sPGA(0) | 0

17. Secondary Outcome: Change From Baseline in Percent of BSA Involvement
Description: as for outcome 7
Time Frame: Baseline, Wk 100; Baseline, Retreatment Wk 192
Population: All participants with Plaque Ps who received at least 1 dose of study drug and had at least 1 post-dose measurement of PASI after study treatment and entered Period 5. Participants with missing BSA at Wks 100 and 192 were imputed by last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: percentage of BSA
Arm/Group | 80 mg Ixekizumab (LY2439821)
Number analyzed (Participants) | 67
percentage of BSA
  Baseline, Wk 100 | -24.7 (17.32)
  Baseline, Wk 192 | -40.2 (21.18)

18. Secondary Outcome: Change From Baseline in NAPSI
Description: The NAPSI is a numeric, reproducible, objective tool for evaluation of fingernail Ps. This scale is used to evaluate the severity of fingernail bed Ps and fingernail matrix Ps by area of involvement in the fingernail unit. The fingernail is divided with imaginary horizontal and longitudinal lines into quadrants. Each fingernail is given a score for fingernail bed Ps 0 (none) to 4 (Ps in 4 quadrants of the fingernail) and fingernail matrix Ps 0 (none) to 4 (Ps in 4 quadrants in matrix), depending on the presence (score of 1) or absence (score of 0) of any of the features of fingernail bed or matrix Ps in each quadrant. The NAPSI score of a fingernail is the sum of scores in fingernail bed and fingernail matrix from each quadrant (maximum of 8). Each fingernail is evaluated, then the sum of all the fingernails equals the total NAPSI score with a range 0 to 80. Higher scores indicate more severe psoriasis.
Time Frame: Baseline, Wk 100; Baseline, Retreatment Wk 192
Population: All participants with Plaque Ps who received at least 1 dose of study drug and had at least 1 post-dose measurement of PASI after study treatment and entered Period 5. Participants with missing NAPSI at Wks 100 and 192 were imputed by LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 80 mg Ixekizumab (LY2439821)
Number analyzed (Participants) | 36
units on a scale
  Baseline, Wk 100 | -16.8 (19.87)
  Baseline, Wk 192 | -21.4 (26.31)

19. Secondary Outcome: Change From Baseline in PSSI
Description: as for outcome 9
Time Frame: Baseline, Wk 100; Baseline, Retreatment Wk 192
Population: All participants with Plaque Ps who received at least 1 dose of study drug and had at least 1 post-dose measurement of PASI after study treatment and entered Period 5. Participants with missing PSSI at Wks 100 and 192 were imputed by LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 80 mg Ixekizumab (LY2439821)
Number analyzed (Participants) | 64
units on a scale
  Baseline, Wk 100 | -8.5 (16.16)
  Baseline, Wk 192 | -23.2 (15.17)

20. Secondary Outcome: Change From Baseline in QIDS-SR16 Score
Description: QIDS-SR16 is a participant-administered, 16-item instrument intended to assess the existence and severity of symptoms of depression. A participant is asked to consider each statement as it relates to the way they have felt for the past 7 days and rate each on a 4-point scale: 0 (best) to 3 (worst) scale. The sum of the 16 items corresponding to 9 depression domains [sad mood, concentration, self-criticism, suicidal ideation, interest, energy/fatigue, sleep disturbance (initial, middle and late insomnia or hypersomnia), decrease/increase in appetite/weight, and psychomotor agitation/retardation] give a single total scores range from 0 to 27, with higher scores indicating greater symptom severity.
Time Frame: Baseline, Wk 100; Baseline, Retreatment Wk 192
Population: All participants with Plaque Ps who received at least 1 dose of study drug and had at least 1 post-dose measurement of PASI after study treatment and entered Period 5. Participants with missing QIDS-SR16 at Wks 100 and 192 were imputed by LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 80 mg Ixekizumab (LY2439821)
Number analyzed (Participants) | 46
units on a scale
  Baseline, Wk 100 | -0.5 (4.02)
  Baseline, Wk 192 | -1.8 (3.87)

21. Secondary Outcome: Change From Baseline in Itch NRS Score
Description: The Itch NRS is a participant-administered, 11-point horizontal scale anchored at 0 (no itch) and 10, (worst itch imaginable). Overall severity of a participant's itching from Ps is indicated by circling the number that best describes the worst level of itching in the past 24 hours.
Time Frame: Baseline, Wk 100; Baseline, Retreatment Wk 192
Population: All participants with Plaque Ps who received at least 1 dose of study drug and had at least 1 post-dose measurement of PASI after study treatment and entered Period 5. Participants with missing Itch NRS at Wks 100 and 192 were imputed by LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 80 mg Ixekizumab (LY2439821)
Number analyzed (Participants) | 67
units on a scale
  Baseline, Wk 100 | -1.1 (2.62)
  Baseline, Wk 192 | -4.9 (2.59)

22. Secondary Outcome: Change From Baseline in DLQI Score
Description: DLQI is a participant-administered, 10-question, validated, quality-of-life questionnaire that covers 6 domains, including symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. Response categories include 0 (not at all), 1 (a little), 2 (a lot), and 3 (very much) and unanswered ("not relevant") responses were scored as "0." Total scores range from 0 to 30, with higher scores indicating greater quality of life impairment. A 5-point increase in total score from baseline is considered clinically relevant.
Time Frame: Baseline, Wk 100; Baseline, Retreatment Wk 192
Population: All participants with Plaque Ps who received at least 1 dose of study drug and had at least 1 post-dose measurement of PASI after study treatment and entered Period 5. Participants with missing DLQI at Wks 100 and 192 were imputed by LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 80 mg Ixekizumab (LY2439821)
Number analyzed (Participants) | 67
units on a scale
  Baseline, Wk 100 | -2.3 (4.83)
  Baseline, Wk 192 | -8.9 (5.70)

23. Secondary Outcome: Change From Baseline in Participants Assessment of Joint Pain VAS
Description: The pain VAS is a participant-administered single-item scale designed to measure current joint pain from PsA using a 100-mm horizontal VAS. Overall severity of participant's joint pain from PsA is indicated by placing a single mark on the horizontal 100-mm scale from 0mm (no pain) to 100 mm (pain as severe as you can imagine).
Time Frame: Baseline, Wk 100; Baseline, Retreatment Wk 192
Population: All participants with Plaque Ps who received at least 1 dose of study drug and had at least 1 post-dose measurement of PASI after study treatment and entered Period 5. Participants with missing Joint Pain VAS at Wks 100 and 192 were imputed by LOCF.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 80 mg Ixekizumab (LY2439821)
Number analyzed (Participants) | 10
mm
  Baseline, Wk 100 | -12.8 (39.59)
  Baseline, Wk 192 | -43.8 (25.66)

24. Secondary Outcome: Number of Participants Achieving ACR20
Description: ACR20 response is defined as ≥20% improvement from baseline for TJC and SJC and in at least 3 of the following 5 criteria: participant's assessment of Joint Pain VAS, Patient's Global Assessment of Disease Activity VAS, Physician's Global Assessment of the Disease Activity VAS, participant's assessment of physical function using the HAQ-DI, or CRP or the ESR.
  Analysis population included participants with PsA who had 3 or more tender joints and 3 or more swollen joints at screening and baseline.
Time Frame: Wk 100 and Wk Retreatment Wk 192
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | 80 mg Ixekizumab (LY2439821)
Number analyzed (Participants) | 10
Participants
  Wk 100 | 0
  Wk 192 | 0

ADVERSE EVENTS:
Description: All enrolled participants.
Groups:
- LY2439821 80mg-Combined Induction and Maintenance Periods; LY2439821 80mg-Drug-Free Period; LY2439821 80mg-Retreatment Period; LY2439821 80mg-Post-Treatment Follow-Up Period: Ixekizumab:
  Period 2 - Participants were administered two 80-mg SC injections at Week 0, followed by 80-mg given as 1 SC injection Q2W (Weeks 2, 4, 6, 8, and 10).
  Period 3 - Participants were administered 80-mg as 1 SC injection Q4W (Week 12 up to Week 52) Period 4 - No ixekizumab administered (drug-free), (Week 52 up to Week 100) Period 5 - Participants who had a Ps relapse during the drug-free period (Period 4) or who completed Period 4 were administered 80 mg as 1 SC injection Q4W for up to 192 weeks.
Arm/Group | LY2439821 80mg-Combined Induction and Maintenance Periods | LY2439821 80mg-Drug-Free Period | LY2439821 80mg-Retreatment Period | LY2439821 80mg-Post-Treatment Follow-Up Period
Serious Adverse Events (participants affected / at risk) | 4/91 | 3/70 | 9/80 | 0/88
Other Adverse Events (participants affected / at risk) | 61/91 | 18/70 | 52/80 | 2/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2439821 80mg-Combined Induction and Maintenance Periods (N=91) | LY2439821 80mg-Drug-Free Period (N=70) | LY2439821 80mg-Retreatment Period (N=80) | LY2439821 80mg-Post-Treatment Follow-Up Period (N=88)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperplastic cholecystopathy (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2439821 80mg-Combined Induction and Maintenance Periods (N=91) | LY2439821 80mg-Drug-Free Period (N=70) | LY2439821 80mg-Retreatment Period (N=80) | LY2439821 80mg-Post-Treatment Follow-Up Period (N=88)
Diarrhoea (Gastrointestinal disorders) | 5 (10) | 1 (1) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 8 (45) | 0 (0) | 2 (7) | 0 (0)
Pyrexia (General disorders) | 2 (8) | 0 (0) | 5 (9) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 7 (8) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 2 (2) | 1 (1) | 5 (5) | 0 (0)
Seasonal allergy (Immune system disorders) | 6 (6) | 0 (0) | 3 (3) | 0 (0)
Folliculitis (Infections and infestations) | 3 (3) | 2 (4) | 7 (7) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 3 (3) | 9 (12) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 36 (48) | 6 (8) | 16 (28) | 0 (0)
Alanine aminotransferase increased (Investigations) | 5 (5) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 2 (2) | 5 (5) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (2) | 6 (6) | 2 (2)
Headache (Nervous system disorders) | 5 (5) | 2 (2) | 3 (3) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1) | 2 (2) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 6 (9) | 0 (0) | 5 (5) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 11 (13) | 1 (1) | 10 (11) | 0 (0)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 9 (9) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0) | 5 (5) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 8 (9) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 8 (8) | 3 (3) | 3 (4) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 7 (7) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days